CLINICAL TRIAL: NCT00582920
Title: Investigation of Changes in Bone Scan Imaging Before and After Intravenous Bisphosphonate Therapy for Osseous Metastases From Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 05-133
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Osseous Lesions From Metastatic Breast Cancer
Keywords: osseous lesions; breast cancer; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Radiation: Zometa™ — Patients who will be receiving zoledronic acid therapy and are scheduled for an extent of disease evaluation with bone scan would undergo a second bone scan within 1 day of zoledronic acid therapy to assess changes in imaging.
  Other Names: Zoledronic acid

SUMMARY:
The purpose of this study is to examine for changes in the bone scan after treating with zoledronic acid (Zometa™). This study is designed to show if intravenous (IV) bisphosphonates, which are infused by vein, such as pamidronate (Aredia™) or zoledronic acid (Zometa™), cause changes in the result of bone scans in women with metastatic breast cancer. Both bone scans and the IV bisphosphonates are components of routine care of women with breast cancer that has spread to the bone.

DETAILED DESCRIPTION:
Presently, intravenous bisphosphonates are routinely used every 3 to 4 weeks in patients with osseous metastases from breast cancer. However, there is no data addressing the effects of intravenous bisphosphonate therapy on the results of bone scan imaging. Therefore, the first step in the collaboration between MSKCC Breast Cancer Medicine Service and Nuclear Medicine Service is to define whether or not intravenous bisphosphonate therapy affects the results of bone imaging with the standard technetium, Tc-99m MDP. Women receiving intravenous bisphosphonate therapy for breast cancer metastases involving bone at MSKCC are eligible for this diagnostic clinical is no therapeutic intent in this study.

Bone Scan performed before intravenous bisphosphonate therapy (baseline as clinically indicated). Ideally, the bone scan will be performed immediately before to, bisphosphonate therapy.

Zoledronic acid, intravenous bisphosphonate therapy (as clinically indicated)

Bone Scan performed within 1 day after intravenous bisphosphonate therapy (study test).

Number of lesions seen in the baseline and study test will be counted and compared for changes in imaging results induced by intravenous bisphosphonate therapy.

The number of lesions detected by bone scan pre and post therapy will be recorded and the difference will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving intravenous biphosphonate therapy (zoledronic acid 4 mg or renal dose equivalent) as part of their treatment regimen, who are diagnosed with metastatic breast cancer involving surrounding bone.
* Patients must have had prior treatment zoledronic acid (4 mg or adjusted dose for renal function) within 8 weeks.
* The patients clinical status as assessed by a treating physician must be deemed appropriate for continuing treatment with zoledronic acid
* The patient's clinical status, as assessed by a treating physician, must be deemed appropriate for an evaluation with a bone scan
* The patient's medical status as assessed by a treating physician must be medically appropriate to receive zoledronic acid within the study time frame and in association with the study bone scan

Exclusion Criteria:

* No evidence of bone metastases, or less than 3 osseous lesions felt to be consistent with bone metastases, on most recent bone scan performed for clinical indications prior to study entry.
* Patients with illnesses, or conditions that would prevent them from understanding the nature of the study and complying with the protocol requirements

Ages: 18 Years to 110 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Evaluate whether routine clinical use of intravenous zoledronic acid therapy affects technetium methylidene diphosphonate (Tc-99 MDP) uptake in bone metastases. | January 2009

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Grewal, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org